CLINICAL TRIAL: NCT03037918
Title: Effect of Yakult Ingestion on Diet-induced Insulin Resistance in Humans. A Large-cohort, Mechanistic Follow-up Study.
Brief Title: Effect of Yakult Ingestion on Diet-induced Insulin Resistance in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Yakult Honsha Co., LTD (Industry)
Responsible Party: Principal Investigator, Carl Hulston, Lecturer in Sports Nutrition, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: R16-P132
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Insulin Sensitivity; Insulin Resistance; Type 2 Diabetes Mellitus
Keywords: Gut Microbiota; High Fat Diets; Probiotics; Glycaemic Control
MeSH Terms: conditions — Insulin Resistance; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Open label, control trial
Masking Description: Participants will be given a unique identifier, which will not disclose the treatment group. All biological samples will be labelled with only the unique identifier.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Participants will receive 2 x 65mL doses of Yakult light per day, for 28 days.
  Participants will consume a high-fat (65% of kilocalories) high-calorie (150% of requirements) diet from day 21 to day 28.
  Interventions: Dietary Supplement: Yakult light
- Control Group (No Intervention): Participants will consume a high-fat (65% of kilocalories) high-calorie (150% of requirements) diet from day 21 to day 28.

INTERVENTIONS:
Dietary Supplement: Yakult light — A fermented milk drink containing the probiotic Lactobacillus casei Shirota
  Arms: Treatment Group

SUMMARY:
Participants will be randomly allocated to either Yakult ingestion or a control group. For the first 20 days, subjects will consume their normal diet (keeping a detailed food diary throughout). On days 21-28 they will switch to a high-fat/high-calorie diet.

The investigators hypothesise that consuming a high-fat, high-energy diet for 7 days will alter the composition of the gut microbiota and induce metabolic endotoxaemia / systemic inflammation as well as decreasing whole body insulin sensitivity (as we have shown previously). In contrast, the investigators hypothesise that consuming Yakult for 21 days before and 7 days throughout the high-fat diet will maintain a favourable gut microbiota and prevent metabolic endotoxaemia / systemic inflammation and thus maintain insulin action / insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged 18-30
* Physically active (exercising at least 3 times per week for more than 30 min at a time)
* Non-smoker
* Free from cardiovascular or metabolic disease
* Weight stable for at least 6 months
* Normal body mass index (BMI: 18.5-24.9 kg/m2)*
* Compliant (i.e. understands and is willing, able and likely to comply with all study requirements)

  * Note: If BMI is >24.9, but body fat % (as measured by bioelectrical impedance analysis) is below 21% in males and 31% in females, then the subject may still be recruited at the PI's discretion.

Exclusion Criteria:

* Using probiotic or prebiotic supplements within the previous 3 months
* Vegetarians and vegans
* Diagnosis of insulin resistance, pre-diabetes or full diabetes
* Underweight (determined as BMI less than 18.5 kg/m2)
* Overweight or obese (determined as BMI greater than 24.9 kg/m2)
* Those on a calorie controlled diet or other dietary restrictions that would prevent them from consuming the probiotic treatment and high fat/high calorie diet.
* Those who are unwilling to restrict their intake of fermented dairy products.
* Those with known or suspected food intolerances, allergies or hypersensitivity
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study.
* Participation in another clinical trial
* Those who have donated blood within 3 months of the screening visit and participants for whom participation in this study would result in having donated more than 1500 ml of blood in the previous 12 months.
* Participants who take any form of regular medication that is known to affect either the gut microbiota and/or insulin sensitivity or who have taken any antibiotics in the previous 3 months.
* Participants who know they would not be available for all the lab visits during the 4-week study period.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2017-02-03 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Whole body insulin sensitivity index | The change between pre- and post-high fat diet (assessed on days 21 and 28)
  Assessed by oral glucose tolerance test.

SECONDARY OUTCOMES:
Body Mass Index | Day 0, Day 21 and Day 28
  Calculated from height and weight.
Fasting plasma glucose concentration | Day 0, Day 21 and Day 28
  Measured in fasting plasma sample.
Fasting serum insulin concentration | Day 0, Day 21 and Day 28
  Measured in fasting serum sample.
Fasting plasma triglyceride concentration | Day 0, Day 21 and Day 28
  Measured in fasting plasma sample.
Metabolic endotoxaemia | Day 0, Day 21 and Day 28
  Plasma markers of endotoxaemia
Markers of systemic inflammation | Day 0, Day 21 and Day 28
  Selected plasma cytokines and chemokines
Incretin response to glucose ingestion | Day 0, Day 21 and Day 28
  GLP-1
Microbiome analysis | Day 0, Day 21 and Day 28
  Faecal DNA analysis of the gut microbiota

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Hulston, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom